CLINICAL TRIAL: NCT00946634
Title: Phase 4 - Ozone Therapy in Endodontic Practice, in Vivo Study
Brief Title: Ozone Therapy in Endodontic Practice, in Vivo Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Carlos Goes Nogales, Master, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 154/06
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Primary Apical Periodontite
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ozone Gas (Experimental): Endodontic protocol preconized by University of Sao Paulo associated to ozone gas 40 mg/L
  Interventions: Drug: Ozone
- Control (Active Comparator): Regular endodontic protocol preconized by University of Sao Paulo
  Interventions: Drug: Control (no last irrigation)
- Aqueous Ozone (Experimental): Endodontic protocol preconized by University of Sao Paulo associated to Aqueous ozone 40mg/L
  Interventions: Drug: Aqueous Ozone

INTERVENTIONS:
Drug: Ozone — Regular endodontic protocol preconized by University of Sao Paulo. Root canal irrigation with 1% Sodium Hypochlorite associated to Endo PTC (10mL), final irrigation with EDTA-T 17% remaining for 3 minutes. After a last foaming with ozone gas (Philozon, Santa Catarina, Brazil) at 40mg/L concentration.
  Other Names: Group 2
  Arms: Ozone Gas
Drug: Control (no last irrigation) — Regular endodontic protocol preconized by University of Sao Paulo. Root canal irrigation with 1% Sodium Hypochlorite associated to Endo PTC (10mL), final irrigation with EDTA-T 17% remaining for 3 minutes.
  Other Names: Group 1
  Arms: Control
Drug: Aqueous Ozone — Regular endodontic protocol preconized by University of Sao Paulo. Root canal irrigation with 1% Sodium Hypochlorite associated to Endo PTC (10mL), final irrigation with EDTA-T 17% remaining for 3 minutes. A last irrigation with 10mL of ozonated water at 40mg/mL concentration
  Other Names: Group 3
  Arms: Aqueous Ozone

SUMMARY:
The ozone therapy has been coming up as a new therapeutic modality. Medicine has been practicing since XIX century and counted great results. It is indicated for the treatment of 260 different pathologies. The researches in Dentistry has showed promising results, indicating a wide spread action in whole dental specialties. The great oxidative power of ozone provides a great antimicrobial effect and it increases the adenosine triphosphate (ATP) synthesis that can be considered as a general improvement of the cell metabolism, which can potentize the repair process. Thus, these facts justify the present study which will assess the increase of speed of apical periodontite repair.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* Radiographic evidence of apical periodontite
* No previous root canal treatment

Exclusion Criteria:

* Unhealthy patients
* Regular response to sensibility test
* Previous root canal treatment

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Acceleration in repair by healing of apical periodontite | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: José L Lage-Marques, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- Fundação para o Desenvolvimento Científico e Tecnológico da Odontologia of University of Sao Paulo, São Paulo, São Paulo, Brazil